CLINICAL TRIAL: NCT04968678
Title: Exploring the Relationship Between Duration of the Amplified P-Wave Arrhythmia and Recurrence in Patients With Persistent, Long Persistent or Paroxysmal AF Undergoing Cryoablation
Brief Title: Exploring P-Wave Duration in Arrhythmia Recurrence in Patients Undergoing AF Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nik Spinthakis (Other)
Collaborators: Dr Guy Haywood (Unknown)
Responsible Party: Sponsor-Investigator, Nik Spinthakis, PI,Cardiology ST5,MBBS,MRCP,MD, University Hospital Plymouth NHS Trust
Organization: University Hospital Plymouth NHS Trust (Other)
Other Study IDs: IRAS 287263-Local21/CAR/492
Record Dates: First submitted 2021-06-26; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation Recurrent
Keywords: P-wave duration; AF; cryoablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: P-wave duration measurement on 12 lead ECG with standard parameters — Hospital records will be used in order to obtain baseline characteristics and the most recent 12-lead ECG in sinus rhythm prior to ablation will be used to calculate PWD. Measurement of the PWD will be obtained at standard surface ECG recording settings of 25mm/s and 10mm/mV and measured accordingly to our previous protocol. In brief, all ECGs obtained will subsequently be anonymised and randomised by an Independent Clinical Investigator (ICI) before measured by the main clinical investigators blinded to initial results. If a dispute of the measurements arouse, consensus will be used to resolve it after consulting the Chief Investigator (CI) blinded to the results. Bland-Altman plots to minimise bias will be used

SUMMARY:
The aim of this study is to investigate whether P-wave duration in a baseline surface 12-lead ECGs correlates with recurrence of AF recurrence post successful ablation at the time of the procedure.

DETAILED DESCRIPTION:
Patients with paroxysmal AF are often treated arrhythmia-free (75%) with a single catheter ablation at 12 months post procedure . In contrast, in patients with persistent AF or long persistent AF, catheter ablation is more complex and often yields in lower success rates of around 50% often requiring multiple attempts .

The success rates remain low despite several different ablation sites having been proposed (additional lines plus PVI, epicardial approach).

There is growing evidence that PWD is associated with the extent of left atrial scarring and this can be used a potential predictor of AF recurrence . Moreover, results from the investigators group has previously shown that PWD correlated with the duration of the AF and this could be altered by extensive ablation .

It is uncertain whether PWD prior to any procedure for persistent AF, long persistent or paroxysmal AF can accurately predict failure of procedure.

This is a single centre observational study of persistent, long persistent and paroxysmal AF population who have undergo AF cryoablation in University Hospital Plymouth . All patients receive this current procedure as standard of care.

This study does not involve any patient contact out of the standard routine clinical follow up and therefore no public involvement has been sought.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent, long persistent or paroxysmal AF undergone AF cryoablation from 2016 onwards
2. Age >18
3. Patient does not meet exclusion criteria -

Exclusion Criteria:

1. Patients whose records cannot be obtained
2. Patients with persistent, long persistent or paroxysmal AF undergone AF ablation prior to 2016
3. Patients with no documented ECG in sinus rhythm prior to ablation
4. Patients not undergoing cryoablation for AF -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective single centre study of the investigators current registry of patients undergoing AF ablation from existing clinical procedural database which contains a record of all cryoablation performed within the hospital.
  All records once obtained from the main database, will then be uploaded into a password protected Excel spreadsheet and anonymised at the time of entry by the ICI.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-01-13 (Estimated); Study Completion 2023-05-13 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation. | 24 months
  Primary.This will be documented in a 12 lead ECG >30sec post ablation according to standard operation procedures follow up. Patients are actively followed up in regular intervals (4-12-24 months) post procedure and are able to contact department for advise if clinically suspected recurrence of atrial fibrillation. This is well studied and documented in previous studies as an outcome of measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To comply with the Data Protection legislation information must be collected and used fairly, stored safely and not disclosed to any unauthorised person. This applies to both manual and electronically held data.
  The Chief Investigator will preserve the confidentiality of participants taking part in the study and ensure the EU General Data Protection Regulation (GDPR) in conjunction with the UK Data Protection Act 2018, which sets out the statutory requirements for the processing of personal data, is adhered to.
  Study documents will be anonymised by allocation of a study number, and will not contain personal identifiable data. Finalised data in an anonymised electronic format will be sent via encrypted USB devices in order to be analysed in a password protected computer. For each patient, a study number will be allocated, and data entered on an anonymised electronic CRF (case report form) in the way of an excel spreadsheet.